CLINICAL TRIAL: NCT01344928
Title: The Effects of Short-time High-intensity Interval Training on Tissue Glucose and Fat Metabolism in Healthy Subjects and Patients With Type 2 Diabetes
Acronym: HITPET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Collaborators: European Foundation for the Study of Diabetes (Other); Ministry of Education and Culture, Finland (Other); Orion Farmos Research Foundation (Unknown); Academy of Finland (Other); Turku PET Centre (Unknown); University of Turku (Other); Verve Research, Oulu, Finland (Other); University of Helsinki (Other)
Responsible Party: Jarna Hannukainen, Turku PET Centre
Other Study IDs: 95/180/2010
Record Dates: First submitted 2011-04-28; First posted 2011-04-29 (Estimated); Last update posted 2011-04-29 (Estimated); Status verified 2011-04

CONDITIONS: Type 2 Diabetes Mellitus; Healthy Volunteers
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HIT training (Experimental)
  Interventions: Behavioral: HIT exercise intervention
- Aerobic exercise training (Active Comparator)
  Interventions: Behavioral: Aerobic exercise intervention

INTERVENTIONS:
Behavioral: HIT exercise intervention
  Arms: HIT training
Behavioral: Aerobic exercise intervention
  Arms: Aerobic exercise training

SUMMARY:
The objectives of this study are to investigate the effects of short-time high-intensity interval training on tissue glucose and fat metabolism in healthy lean subjects and type 2 diabetic patients using modern and noninvasive imaging methods positron emission tomography (PET), magnetic resonance imaging (MRI) and magnetic resonance spectroscopy (MRS).

ELIGIBILITY:
Inclusion Criteria:

The healthy patients

1. Age 40-55
2. BMI 18.5-30
3. Fasting plasma glucose less than 6.1 mmol/l
4. Normal glucose tolerance test (OGTT)

The type 2 diabetic patients:

1. Age-, sex-, and BMI-matched with the study subjects in the phase 1
2. In a good treatment balance
3. Glycated haemoglobin (HbA1c) less than 7.5 mmol/l
4. Two hours glucose value in oral glucose tolerance test (OGTT) less than 10.0 mmol/l

Exclusion Criteria:

The healthy patients

1. Blood pressure > 140/90 mmHg
2. Any chronic disease
3. Any chronic medical defect or injury which hinder/interfere everyday life
4. History of anorexia nervosa or bulimia
5. History of rest or exercise-induced asthma
6. Previous use of anabolic steroids, additives or any other substrates
7. Smoking of tobacco, taking of snuffs, or use of narcotics.
8. Significant use of alcohol
9. Any other condition that in the opinion of the investigator could create a hazard to the subject safety, endanger the study procedures or interfere with the interpretation of study results
10. Presence of any ferromagnetic objects that would make MR imaging contraindicated
11. Current or history of regular and systematic exercise training
12. VO2max >40 ml/min/kg

The type 2 diabetic patients:

1. Any other chronic disease than diabetes
2. Blood pressure > 140/90 mmHg
3. Any chronic medical defect or injury which hinder/interfere everyday life
4. History of anorexia nervosa or bulimia
5. History of rest or exercise-induced asthma
6. Smoking of tobacco, taking of snuffs, or use of narcotics.
7. Any other condition that in the opinion of the investigator could create a hazard to the subject safety, endanger the study procedures or interfere with the interpretation of study results
8. Presence of any ferromagnetic objects that would make MRI imaging contraindicated
9. Current or history of regular and systematic exercise training
10. VO2max >40 ml/ min/kg

Ages: 40 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Turku PET Centre, Turku, Finland

REFERENCES:
- [Derived] Ojala R, Motiani KK, Ivaska KK, Arponen M, Eskelinen JJ, Virtanen KA, Loyttyniemi E, Heiskanen MA, U-Din M, Nuutila P, Kalliokoski KK, Hannukainen JC. Bone Marrow Metabolism Is Impaired in Insulin Resistance and Improves After Exercise Training. J Clin Endocrinol Metab. 2020 Dec 1;105(12):e4290-303. doi: 10.1210/clinem/dgaa516. PMID 32785654
- [Derived] Motiani KK, Collado MC, Eskelinen JJ, Virtanen KA, Loyttyniemi E, Salminen S, Nuutila P, Kalliokoski KK, Hannukainen JC. Exercise Training Modulates Gut Microbiota Profile and Improves Endotoxemia. Med Sci Sports Exerc. 2020 Jan;52(1):94-104. doi: 10.1249/MSS.0000000000002112. PMID 31425383
- [Derived] Heiskanen MA, Motiani KK, Mari A, Saunavaara V, Eskelinen JJ, Virtanen KA, Koivumaki M, Loyttyniemi E, Nuutila P, Kalliokoski KK, Hannukainen JC. Exercise training decreases pancreatic fat content and improves beta cell function regardless of baseline glucose tolerance: a randomised controlled trial. Diabetologia. 2018 Aug;61(8):1817-1828. doi: 10.1007/s00125-018-4627-x. Epub 2018 May 2. PMID 29717337